CLINICAL TRIAL: NCT03809910
Title: An Exploratory, Randomized, Single Center, Partial Crossover, Clinical Study to Evaluate the Dental Plaque Removal Ability of a Prototype Power Toothbrush Versus a Manual Toothbrush After a Single Tooth Brushing Event
Brief Title: Dental Plaque Removal Ability of Prototype Power Toothbrush Versus a Manual Toothbrush in Healthy Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 208112
Record Dates: First submitted 2019-01-07; First posted 2019-01-18 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Dental Plaque
Keywords: Oral Health, Dental care, Lifestyle
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prototype PTB (Gum line mode) (Experimental): Participants will brush their teeth with prototype power toothbrush in Gum line mode with a fluoride toothpaste
  Interventions: Device: Prototype PTB (Gum line mode)
- Prototype PTB (Combined mode) (Experimental): Participants will brush their teeth with prototype power toothbrush in "Gum line" mode with a fluoride toothpaste. Following this, participants will brush their teeth with prototype power toothbrush in 'Interdental' mode with a fluoride toothpaste.
  Interventions: Device: Prototype PTB (Combined mode)
- Reference MTB (Sham Comparator): Participants will brush their teeth with manual toothbrush and fluoride toothpaste.
  Interventions: Device: Reference MTB
- Reference PTB (Active Comparator): Participants will brush their teeth with reference power toothbrush and fluoride toothpaste.
  Interventions: Device: Reference PTB

INTERVENTIONS:
Device: Reference MTB — Participants will brush their teeth with manual toothbrush and 1.3 g ± 0.1 g of fluoride toothpaste (containing 0.76% w/w sodium monofluorophosphate) for 1-timed minute under supervision of study staff.
  Arms: Reference MTB
Device: Reference PTB — Participants will brush their teeth with power toothbrush and 1.3 g ± 0.1 g of fluoride toothpaste (containing 0.76% w/w sodium monofluorophosphate) for 2-timed minute under supervision of study staff.
  Arms: Reference PTB
Device: Prototype PTB (Gum line mode) — Participants will brush their teeth with prototype PTB toothbrush and 1.3 g ± 0.1 g of fluoride toothpaste (containing 0.76% w/w sodium monofluorophosphate) for 2-timed minute in "Gum Line" mode under supervision of study staff.
  Arms: Prototype PTB (Gum line mode)
Device: Prototype PTB (Combined mode) — Participants will brush their teeth with prototype PTB toothbrush and 1.3 g ± 0.1 g of fluoride toothpaste (containing 0.76% w/w sodium monofluorophosphate) for 2-timed minute in "Gum Line" mode and 1-timed minute in "Interdental" mode under supervision of study staff.
  Arms: Prototype PTB (Combined mode)

SUMMARY:
The aim of this study is to evaluate the ability of a prototype power toothbrush (PTB) versus a manual toothbrush in healthy, right-handed manual toothbrush (MTB) participants with no signs of periodontal disease or excessive recession to remove dental plaque after a single tooth brushing event. Prior to each treatment visit, participants will abstain from oral hygiene for a period of 12 hours preceding a pre-brushing dental plaque evaluation. Participants will then brush once under supervision for 2 minutes in 'Gum line' mode and 1-minute in 'Interdental' mode after which re-disclosing and a post-brushing plaque assessment will be carried out.

DETAILED DESCRIPTION:
This study is an exploratory, randomized, single center, 4-treatment, 3-period, partial crossover study in healthy participants with no signs of periodontal disease or excessive recession, to assess a prototype PTB in removing dental plaque after a single brushing event.

At the screening visit, following provision of written informed consent, participants will be provided PTB training to familiarize themselves with how the different modes and different PTBs operate. Eligible participants will be provided with a washout fluoride toothpaste and toothbrush for use at home during the study.

Participants will then be scheduled to attend appointment after a minimum of 3 days. For each treatment visit, participants must abstain from oral hygiene for a period of 12hours, immediately preceding the pre-brushing dental plaque evaluation.

All the participants will undergo an oral soft tissue (OST) examination followed by plaque disclosing and a pre-brushing dental plaque assessment using the Rustogi Modified Navy Plaque Index (RMNPI) index. In in periods 1 and 2, participants will be randomized to the study treatment sequence with the prototype PTB and MTB used in a crossover manner and participants will then brush under supervision followed by disclosing and post-brushing plaque assessments. Participants assigned to the prototype PTB, it will be used for 2 minutes in 'Gum line' mode brushing and 1-minute brushing in 'Interdental' mode.

Participants will then brush once (1.3 grams [g] ± 0.1 g of assigned toothpaste), under supervision of study staff after which disclosing, and a post-brushing plaque assessment will be carried out.

Participants will be allowed to brush with the washout paste following the post assessment plaque assessments. A minimum of three days washout period will follow each treatment period during which period Participants will brush with a standard washout toothpaste

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all the following inclusion criteria to be eligible for enrollment into the study:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is male or female who, at the time of screening, is between the ages of 18 and 65 years, inclusive.
* A participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* A participant that successfully completes the investigational device training visit, understands and is willing to follow product usage instructions, in the opinion of the investigator or designee.
* A participant in good general and mental health, in the opinion of the investigator or medically qualified designee; no clinically significant and relevant abnormalities in medical history or upon oral examination.
* A participant with good dental health based on medical history and oral soft tissue examination at screening.
* A participant with a minimum of 20 permanent gradable teeth (gradable teeth are those where restorative materials cover less than 25% of the tooth surface graded).
* For continued eligibility after the Screening visit, a participant must have a mean RMNPI whole mouth plaque score of ≥ 0.6 at Visit 2, 3, 4 and 5.
* A participant that regularly uses a manual toothbrush in their daily oral hygiene routine.
* A participant that regularly brushes their teeth with their right hand.

Exclusion Criteria:

An individual who meets any of the following exclusion criteria will not be eligible for enrollment into the study:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is a pregnant female (evidenced by positive urine pregnancy test).
* A participant who is a breastfeeding female.
* A male participant able to father children or female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for 5 days after the last assigned treatment.
* A female participant who is of childbearing potential and are sexually active and at risk for pregnancy must agree to use a highly effective method of contraception consistently and correctly for the duration of the active study period and for 5 days after the last assigned treatment.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A participant unwilling or unable to comply with the following Lifestyle Considerations: a) Participants will be requested not to have any elective dental procedures including teeth professionally cleaned, excluding emergency dental treatment ; b)Participants will be requested not to have whitening treatment (including professional or at home use) during the duration of the study; c) Participants will not be permitted to use any other oral care products (i.e. oral rinses, tongue cleaners, whitening, bleaching products) besides the products supplied for this study; d) Eligible participants will be asked to stop using their regular dentifrice and toothbrush from the Screening visit for the duration of the study; e) Participants should abstain from interproximal cleaning (i.e. dental floss, oral irrigators, interdental brushes) for the duration of the study. Participants will be permitted to use toothpicks or floss to remove impacted food only ; f) Prior to Visit 2, 3 and 4:Participants should abstain from all oral hygiene procedures for at least12 hours prior to the scheduled time of their Visit 2, 3 and 4 appointments; g ) On study visit days (Visits 2, 3 and 4) participants must abstain from all food and drink (except water) at least 4 hours prior to their scheduled visits until all measurements have been taken. Water is permitted until 1 hour prior to investigational product administration; h) Participants must abstain from chewing gum and consuming confectionary containing xylitol (e.g. mints) at least 4 hours prior to their scheduled visit; i) On study visit days (Visits 2, 3 and 4) participants must abstain from all alcohol until all measurements have been taken; j) Participants will abstain from caffeine-containing products for at least 4 hours prior to their scheduled Visit 2, 3 and 4 until all measurements have been take; k) Participant will abstain from smoking, chewing tobacco, or smoking E-cigarettes throughout the study.
* A participant who has received a dental prophylaxis within 4 weeks of Screening visit.
* A participant who has received teeth bleaching/whitening (including professional or at home use) within 8 weeks prior to Screening visit.
* A participant who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
* A participant who has received orthodontic therapy or scaling or root planning within 3 months of Screening.
* A participant with high levels of extrinsic stain or calculus deposits which might interfere with dental plaque assessments.
* A participant that has current active caries, excessive gingival recession, severe gingivitis or periodontitis that may, in the opinion of the investigator, compromise the study or the oral health of the participant if they participate in the study.
* A participant with the presence of oral or peri-oral ulceration including herpetic lesions at the time of screening.
* A participant who is at risk of spasms.
* A participant with restorations in a poor state of repair that may, in the opinion of the investigator, compromise the study or the oral health of the participant if they participate in the study.
* A participant with the presence of orthodontic bands or appliances, extensive crowns, partial or full dentures, or fixed retainers on the maxillary or mandibular teeth.
* A participant with a tongue or lip piercing, or any other oral feature that could interfere with the usage of the toothbrush.
* A participant who has used antibiotic treatment within 14 days prior to Screening visit.
* A participant with diagnosed xerostomia or taking any medication that in view of the investigator causes xerostomia.
* A participant with any electronic medical devices (such as pacemakers).
* A participant that has used a chlorhexidine mouthwash within 14 days of Screening visit or used any oral care product that under the criteria of the principal investigator could interfere with dental plaque formation.
* A participant unwilling to abstain from using other oral care products besides those assigned to them in the study.
* A participant with a recent history (within past year) of alcohol or other substance abuse.
* A participant that smokes or uses chew tobacco, or regularly smokes E-cigarettes.
* A participant who has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Mississauga, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in Canada. A total of 40 participants were screened, of whom 39 were randomized for treatment and 1 withdrew consent prior to randomization.
Pre-assignment Details: Participants received 4 treatments in 3 periods: 1. Prototype power toothbrush (PTB) in 'Gumline' mode, 2. Prototype PTB in 'Combined' mode ('Gumline' mode followed by 'Interdental' mode), 3. Reference manual toothbrush (MTB), 4. Reference PTB
Groups:
- Sequence A-B-C: Participants randomized to this group brushed their teeth as follows in supervision of study staff during site visit: Prototype PTB (A) in Period 1 (for 2 timed minutes [min] in 'Gumline' mode and 1 timed min in 'Interdental' mode) followed by Reference MTB (B) in Period 2 (for 1 timed min) and Reference PTB (C) in Period 3 (for 2 timed min). Clinical assessments were performed after 'Gumline' mode and 'Interdental' mode in same treatment period. Each treatment period was followed by a minimum of 3-days washout period and prior to each site visit, participants abstained from all oral hygiene for at least 12 hours. Participants received a fluoride toothpaste and manual toothbrush to use at home during washout period, recorded each brushing occasion (at home) and time of their last brushing prior to their next scheduled appointment on their diary. Overall study duration from first subject first visit (FSFV) to last subject last visit (LSLV) was 32 days.
- Sequence B-A-C: Participants randomized to this group brushed their teeth as follows in supervision of study staff during site visit: Reference MTB (B) in Period 1 (for 1 timed minute) followed by Prototype PTB (A) in Period 2 (for 2 timed minutes in 'Gumline' mode and 1 timed minute in 'Interdental' mode) and Reference PTB in Period 3 (C) (for 2 timed minutes). Clinical assessments were performed after 'Gumline' mode and after 'Interdental' mode in same treatment period. Each treatment period was followed by a minimum of 3-days washout period and prior to each site visit, participants abstained from all oral hygiene for at least 12 hours. Participants received a fluoride toothpaste and manual toothbrush to use at home during the washout period and recorded each brushing occasion (at home) and time of their last brushing prior to their next scheduled appointment on their diary. Overall study duration from FSFV to LSLV was 32 days.
Period: Period 1 (Visit 2)
Arm/Group | Sequence A-B-C | Sequence B-A-C
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0
Period: Washout Period 1 (3 Days)
Arm/Group | Sequence A-B-C | Sequence B-A-C
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0
Period: Period 2 (Visit 3)
Arm/Group | Sequence A-B-C | Sequence B-A-C
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0
Period: Washout Period 2 (3 Days)
Arm/Group | Sequence A-B-C | Sequence B-A-C
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0
Period: Period 3 (Visit 4)
Arm/Group | Sequence A-B-C | Sequence B-A-C
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (m-ITT) population included all participants who are randomized, received at least one of the study treatments and provide at least one post-brushing assessment of efficacy.
Groups:
- All Treatment Combined: All randomized participants received treatment in either sequence A-B-C or sequence B-A-C. Participants in the product sequence A-B-C applied Prototype PTB (A) in Period 1 followed by Reference MTB (B) in Period 2 and Reference PTB (C) in Period 3, whereas, in product sequence B-A-C participants applied Reference MTB (B) in Period 1 followed by Prototype PTB (A) in Period 2 and Reference PTB (C) in Period 3.
Arm/Group | All Treatment Combined
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Whole Mouth Rustogi Modified Navy Plaque Index (RMNPI) Score From Pre-Brushing to Post-Brushing (When Prototype Power Toothbrush [PTB] Was Used in 'Gumline' Mode vs a Reference Manual Toothbrush [MTB])
Description: Change in plaque removal efficacy from pre-brushing to post-brushing in whole mouth (sites A to I) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' mode versus a reference MTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 2 minutes of brushing
Population: Modified Intent-to-Treat (mITT) Population included all randomized participants who had received at least one dose of study products (supervised brushing in study period 1, 2 or 3) and had provided at least one post-brushing assessment of efficacy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Prototype PTB "Gumline": Participants randomized to receive Prototype PTB either in Treatment Period 1 or Treatment Period 2 for 2 timed minutes in 'Gumline' mode. Clinical assessments were performed after the 'Gumline' mode.
- Reference MTB: Participants randomized to receive Reference MTB either in Treatment Period 1 or Treatment Period 2 for 1 timed minute.
Arm/Group | Prototype PTB "Gumline" | Reference MTB
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.38 (0.086) | -0.32 (0.083)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Reference MTB; Test type: Superiority; p < .0001, ANCOVA — Analysis was performed using ANCOVA model with product, sequence as fixed effects, participant as a random effect and two baseline terms as covariates;1-participant-level baseline score,2-period level baseline minus the participant-level baseline; Adjusted Mean Difference = -0.06, 95% CI 2-sided [-0.09 to -0.04], Standard Error of Mean 0.014

2. Secondary Outcome: Change in Marginal RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Gumline' Mode vs a Reference MTB)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing at the gum line (referred as marginal score-sites A to C) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' mode versus a reference MTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 2 minutes of brushing
Population: mITT Population included all randomized participants who had received at least one dose of study products (supervised brushing in study period 1, 2 or 3) and had provided at least one post-brushing assessment of efficacy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Gumline" | Reference MTB
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.50 (0.156) | -0.38 (0.166)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Reference MTB; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.12, 95% CI 2-sided [-0.17 to -0.07], Standard Error of Mean 0.025

3. Secondary Outcome: Change in Proximal RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Gumline' Mode vs a Reference MTB)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing at the proximal tooth areas (referred to as proximal score-sites D and F) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' mode versus a reference MTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 2 minutes of brushing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Gumline" | Reference MTB
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.66 (0.175) | -0.55 (0.140)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Reference MTB; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.11, 95% CI 2-sided [-0.16 to -0.06], Standard Error of Mean 0.025

4. Secondary Outcome: Change in Whole Mouth RMNPI Score From Pre-brushing to Post-brushing (When Prototype PTB Was Used in 'Combined' Mode vs a Reference MTB)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing in whole mouth (site A to I) was assessed using RMNPI score, when prototype PTB used in the 'Combined' Mode ('Gumline' mode followed by 'Interdental' mode) versus a reference MTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: mITT Population included all randomized participants who had received at least one dose of study products (supervised brushing in study period 1, 2 or 3) and had provided at least one post-brushing assessment of efficacy. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Prototype PTB "Combined": Participants randomized to receive Prototype PTB either in Treatment Period 1 or Treatment Period 2 for 2 timed minutes in 'Gumline' mode and 1 timed minute in 'Interdental' mode. Clinical assessments were performed after the 'Gumline' mode and after the 'Interdental' mode.
Arm/Group | Prototype PTB "Combined" | Reference MTB
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.54 (0.054) | -0.32 (0.083)
Statistical Analysis 1: Comparison: Prototype PTB "Combined" vs Reference MTB; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.22, 95% CI 2-sided [-0.25 to -0.19], Standard Error of Mean 0.014

5. Secondary Outcome: Change in Marginal RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Combined' Mode vs a Reference MTB)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing at the gum line (referred as marginal score-sites A to C) was assessed using RMNPI score, when prototype PTB used in the 'Combined' Mode ('Gumline' mode for 2 minutes followed by 'Interdental' mode for 1 minute) versus a reference MTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Combined" | Reference MTB
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.76 (0.141) | -0.38 (0.166)
Statistical Analysis 1: Comparison: Prototype PTB "Combined" vs Reference MTB; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.38, 95% CI 2-sided [-0.43 to -0.33], Standard Error of Mean 0.025

6. Secondary Outcome: Change in Proximal RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Combined' Mode vs a Reference MTB)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing at the proximal tooth areas (referred to as proximal score-sites D and F) was assessed using RMNPI score, when prototype PTB used in the 'Combined' Mode ('Gumline' mode for 2 minutes followed by 'Interdental' mode for 1 minute) versus a reference MTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Combined" | Reference MTB
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.90 (0.106) | -0.55 (0.140)
Statistical Analysis 1: Comparison: Prototype PTB "Combined" vs Reference MTB; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.34, 95% CI 2-sided [-0.39 to -0.29], Standard Error of Mean 0.025

7. Secondary Outcome: Change in Whole Mouth RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Gumline' Mode vs 'Combined' Mode)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing in whole mouth (site A to I) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' mode versus prototype PTB used in the 'Combined' Mode ('Gumline' mode for 2 minutes followed by 'Interdental' mode for 1 minute) after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Gumline" | Prototype PTB "Combined"
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.38 (0.086) | -0.54 (0.054)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Prototype PTB "Combined"; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = 0.15, 95% CI 2-sided [0.13 to 0.18], Standard Error of Mean 0.014

8. Secondary Outcome: Change in Marginal RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Gumline' Mode vs 'Combined' Mode)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing at the gum line (referred as marginal score-sites A to C) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' mode versus prototype PTB used in the 'Combined' Mode ('Gumline' mode for 2 minutes followed by 'Interdental' mode for 1 minute) after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Gumline" | Prototype PTB "Combined"
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.50 (0.156) | -0.76 (0.141)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Prototype PTB "Combined"; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = 0.26, 95% CI 2-sided [0.21 to 0.31], Standard Error of Mean 0.025

9. Secondary Outcome: Change in Proximal RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Gumline' Mode vs 'Combined' Mode)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing at the proximal tooth areas (referred to as proximal score-sites D and F) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' mode versus prototype PTB used in the 'Combined' Mode ('Gumline' mode for 2 minutes followed by 'Interdental' mode for 1 minute) after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assigned on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Gumline" | Prototype PTB "Combined"
Number analyzed (Participants) | 39 | 39
Score on a scale | -0.66 (0.175) | -0.90 (0.106)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Prototype PTB "Combined"; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = 0.23, 95% CI 2-sided [0.18 to 0.28], Standard Error of Mean 0.025

10. Secondary Outcome: Change in Whole Mouth RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Gumline' and 'Combined' Modes Versus a Reference PTB)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing in whole mouth (site A to I) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' and 'Combined' mode versus a reference PTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Reference PTB: Participants randomized to receive Reference PTB in Treatment Period 3 for 2 timed minute.
Arm/Group | Prototype PTB "Gumline" | Prototype PTB "Combined" | Reference PTB
Number analyzed (Participants) | 39 | 39 | 39
Score on a scale | -0.38 (0.086) | -0.54 (0.054) | -0.50 (0.061)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Reference PTB; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = 0.12, 95% CI 2-sided [0.09 to 0.15], Standard Error of Mean 0.014
Statistical Analysis 2: Comparison: Prototype PTB "Combined" vs Reference PTB; Test type: Superiority; p = 0.0214, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.03, 95% CI 2-sided [-0.06 to -0.00], Standard Error of Mean 0.014

11. Secondary Outcome: Change in Marginal RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Gumline' and 'Combined' Modes Versus a Reference PTB)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing at the gum line (referred as marginal score-sites A to C) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' and 'Combined' mode versus a reference PTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Gumline" | Prototype PTB "Combined" | Reference PTB
Number analyzed (Participants) | 39 | 39 | 39
Score on a scale | -0.50 (0.156) | -0.76 (0.141) | -0.67 (0.102)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Reference PTB; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = 0.18, 95% CI 2-sided [0.13 to 0.23], Standard Error of Mean 0.025
Statistical Analysis 2: Comparison: Prototype PTB "Combined" vs Reference PTB; Test type: Superiority; p = 0.0010, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.09, 95% CI 2-sided [-0.14 to -0.04], Standard Error of Mean 0.025

12. Secondary Outcome: Change in Proximal RMNPI Score From Pre-Brushing to Post-Brushing (When Prototype PTB Was Used in 'Gumline' and 'Combined' Modes Versus a Reference PTB)
Description: Change in plaque removal efficacy from pre-brushing to post-brushing at the proximal tooth areas (referred to as proximal score-sites D and F) was assessed using RMNPI score, when prototype PTB used in the 'Gumline' and 'Combined' mode versus a reference PTB after a single brushing event. Dental plaque was assessed on all teeth excluding third molars (Universal Numbering System teeth 2 to 15, and 18 to 31), crowns, and surfaces with cervical restorations for a maximum of 28 eligible teeth. Plaque was assessed on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth; where lower score represents the better plaque removal efficacy. Change from pre-brushing = (post-brushing score - pre-brushing score).
Time Frame: After 3 minutes of brushing
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prototype PTB "Gumline" | Prototype PTB "Combined" | Reference PTB
Number analyzed (Participants) | 39 | 39 | 39
Score on a scale | -0.66 (0.175) | -0.90 (0.106) | -0.86 (0.095)
Statistical Analysis 1: Comparison: Prototype PTB "Gumline" vs Reference PTB; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = 0.20, 95% CI 2-sided [0.15 to 0.25], Standard Error of Mean 0.025
Statistical Analysis 2: Comparison: Prototype PTB "Combined" vs Reference PTB; Test type: Superiority; p = 0.1652, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted Mean Difference = -0.04, 95% CI 2-sided [-0.09 to 0.01], Standard Error of Mean 0.026

ADVERSE EVENTS:
Time Frame: 37 Days
Description: Safety population: all participants who were eligible to participate in the study and had participated in the Supervised PTB Training. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported. A participant with multiple occurrences of AEs counted once in AE category. A participant with multiple AEs within a primary system organ class was counted once in system organ class.
Groups:
- Prototype PTB (A): Participants randomized to receive Prototype PTB either in Treatment Period 1 or Treatment Period 2 for 2 timed minutes in 'Gumline' mode and 1 timed minute in 'Interdental' mode. Clinical assessments were performed after the 'Gumline' mode and after the 'Interdental' mode in same treatment period.
- Reference MTB (B): Participants randomized to receive Reference MTB either in Treatment Period 1 or Treatment Period 2 for 1 timed minute.
- Reference PTB (C): Participants randomized to receive Reference PTB in Treatment Period 3 for 2 timed minute.
Arm/Group | Prototype PTB (A) | Reference MTB (B) | Reference PTB (C)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03809910/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03809910/SAP_001.pdf